CLINICAL TRIAL: NCT01348685
Title: Effect of Drinking Liquid Compared to Eating Solid Treatment of Sugars or Whey Protein on Short-term Appetite and Food Intake
Brief Title: Comparing Liquid Versus Solid Forms of Sugars and Whey Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Mondelēz International, Inc. (Industry); Canadian Sugar Institute (Unknown)
Responsible Party: Dr. G. Harvey Anderson, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Solid and liquid 1
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Compare the effect of solid vs. liquid forms of sugars on satiety and food intake
Other: the effect of solid vs. liquid forms of gelatin on appetite and food intake
Other: The effect of solid vs. liquid forms of whey protein on food intake

SUMMARY:
To compare the effect of eating solid vs. drinking liquid forms of gelatin, sucrose and its component mixtures and whey protein on subjective appetite and food intake in young men.

DETAILED DESCRIPTION:
Three randomized cross-over design experiments were used to compare the effect of solid and liquid forms of gelatin (6 g) in experiment 1, sucrose (75 g) and a mixture of 50% glucose/ 50% fructose (G50:F50) in experiment 2, and acid and sweet whey protein (50 g) in experiment 3 on healthy normal weight males . The controls were water (experiment 1 and 3) and calorie-free sweetened water with gelatin (sweet gelatin, experiment 1) or without gelatin (sweet control, experiment 2). Subjective average appetite was measured by visual analogue scales frequently over 1 h and ad libitum food intake was measured 1 h after the treatment consumptions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lean males with BMI between 18- 24.9 kg/m2 and an age range of 19 to 28 years were recruited for the three experiments.

Exclusion Criteria:

* Diabetics (fasting blood glucose ≥ 7.0 mmol/L), smokers, breakfast skippers or dieters were excluded from the experiments. Individuals under medications or with a history of liver or kidney disease and major medical or surgical event within the last six months were excluded.

Ages: 19 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
subjective appetite and short term food intake | 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Department of Nutritional Sciences, Toronto, Ontario, Canada